CLINICAL TRIAL: NCT00376948
Title: Phase II Trial of Novasoy®, Gemcitabine, and Erlotinib in Locally Advanced or Metastatic Pancreatic Cancer
Brief Title: Genistein, Gemcitabine, and Erlotinib in Treating Patients With Locally Advanced or Metastatic Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000495776; P30CA022453 (NIH); WSU-2005-006; WSU-025806MP4F
Record Dates: First submitted 2006-09-13; First posted 2006-09-15 (Estimated); Results first posted 2014-08-26 (Estimated); Last update posted 2021-03-01 (Actual); Status verified 2021-02

CONDITIONS: Pancreatic Cancer
Keywords: adenocarcinoma of the pancreas; stage III pancreatic cancer; stage IV pancreatic cancer; recurrent pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Genistein; Erlotinib Hydrochloride; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Novasoy®, Gemcitabine & Erlotinib (Experimental): Novasoy® 396 mg (177 mg of Isoflavones) twice-daily starting daay -7 until day 28; Gemcitabine 1000 mg/m2 days 1, 8, & 15; Erlotinib 150 mg day 1 until day 28
  Interventions: Dietary Supplement: genistein; Drug: erlotinib hydrochloride; Drug: gemcitabine hydrochloride

INTERVENTIONS:
Dietary Supplement: genistein
Drug: erlotinib hydrochloride
Drug: gemcitabine hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as gemcitabine, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Erlotinib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Genistein may help gemcitabine and erlotinib kill more tumor cells by making tumor cells more sensitive to the drugs.

PURPOSE: This phase II trial is studying how well giving genistein together with gemcitabine and erlotinib works in treating patients with locally advanced or metastatic pancreatic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the 6-month survival rate of patients with locally advanced or metastatic pancreatic cancer treated with genistein, gemcitabine hydrochloride, and erlotinib hydrochloride.

Secondary

* Determine the frequency of objective tumor response rate in these patients.
* Determine the time to treatment failure in these patients.
* Determine the effect of baseline expression of pAKT and activation of NF-kappaB on survival of patients treated with this regimen.
* Determine the overall time to disease progression in these patients.
* Estimate the quantitative and qualitative toxicities of this regimen in these patients.

OUTLINE: This is a multicenter study.

Patients receive oral genistein twice daily on days -7 to 28 in course 1 and on days 1-28 in all other courses. Patients also receive gemcitabine hydrochloride IV over 30 minutes on days 1, 8, and 15 and oral erlotinib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed pancreatic adenocarcinoma

  * Locally advanced or metastatic disease by radiological evidence
* Must have biopsy material consisting of 10 unstained slides or paraffin-embedded tissue blocks available for correlative studies
* No endocrine tumor or lymphoma of the pancreas
* No history of CNS (central nervous system) metastases

PATIENT CHARACTERISTICS:

* SWOG (Southwest Oncology Group) performance status 0-1
* Life expectancy ≥ 12 weeks
* Platelet count ≥ 100,000/mm^3
* Absolute neutrophil count ≥ 1,500/mm^3
* Bilirubin < 2.0 mg/dL
* AST (aspartate aminotransferase) and ALT (alanine aminotransferase) < 1.5 times upper limit of normal
* Creatinine < 1.5 mg/dL
* Albumin > 2.5 g/dL
* INR (international normalized ratio) < 1.3 (in the absence of ongoing treatment with warfarin)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No active infection
* No condition that would limit the ability to receive oral medications
* No requirement for a gastrostomy tube for the administration of drugs
* No serious concurrent systemic disorder, that, in the opinion of the investigator, is incompatible with the study
* No active second primary malignancy within the past year except in situ carcinoma of the cervix or adequately treated basal cell carcinoma of the skin
* No allergy to any study drug

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy for metastatic disease

  * Prior adjuvant chemotherapy allowed provided it was completed at least 6 months ago
* No prior gemcitabine hydrochloride or epidermal growth factor receptor-inhibiting agents
* No other concurrent chemotherapy, immunotherapy, tumor-directed hormonal therapy, or radiotherapy
* No other concurrent investigational agents
* No other concurrent antitumor therapy

Ages: 21 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2005-05; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Khaldoun Almhanna, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute; Fazlul H. Sarkar, PhD, Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - M. D. Anderson Cancer Center at University of Texas, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- Novasoy®, Gemcitabine & Erlotinib: Novasoy® 396 mg (177 mg of Isoflavones) twice-daily starting daay -7 until day 28; Gemcitabine 1000 mg/m2 days 1, 8, & 15; Erlotinib 150 mg day 1 until day 28
  genistein
  erlotinib hydrochloride
  gemcitabine hydrochloride
Period: Overall Study
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Started | 20
Completed | 20
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 20
Age, Continuous [Median (Full Range); unit: years] | 58.5 [39 to 75]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 12
Region of Enrollment [Number; unit: participants]
  United States | 20

OUTCOME MEASURES:

1. Primary Outcome: Patients Alive
Time Frame: at 6 months
Measure: Number; unit: participants
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 20
participants | 10

2. Primary Outcome: Median Overall Survival Estimate
Time Frame: up to 17 months
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 20
months | 6.3 [4.6 to 12.6]

3. Secondary Outcome: Overall Objective Response Rate (Complete and Partial Response)
Description: Imaging tests (CT scan, CXR [Chest X-Ray], MRI or imaging studies as clinically indicated
Time Frame: Every 8 weeks
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 18
proportion of patients | 0.056 [0.012 to 0.215]

4. Secondary Outcome: Response Duration
Description: Imaging tests (CT scan, CXR, MRI or imaging studies as clinically indicated). Progressive disesase is defined as a greater than 20% increase in the sum of the longest diameter of target lesions taking as reference the smalles sum of the longest diameter recorded since the treatment started or the appearance of new lesions. Partial response is defined as greater than or equal to 30% reduction in the sum of the longest diameteres of target lesions, taking as reference the baseline sum of the longest diameters.
Time Frame: Every 8 weeks
Measure: Number; unit: days
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 1
days | 73

5. Secondary Outcome: Time to Treatment Failure
Description: Imaging tests (CT scan, CXR, MRI or imaging studies as clinically indicated). Progressive disesase is defined as a greater than 20% increase in the sum of the longest diameter of target lesions taking as reference the smalles sum of the longest diameter recorded since the treatment started or the appearance of new lesions.
Time Frame: Every 8 weeks
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 17
months | 2.04 [1.74 to 3.48]

6. Secondary Outcome: Time to Progression
Description: as for outcome 5
Time Frame: Every 8 weeks
Measure: Median (90% Confidence Interval); unit: moths
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 19
moths | 2.07 [2.04 to 8.34]

7. Secondary Outcome: Grade 3 or Higher Toxicity Evaluation
Description: Toxicity evaluation using NCI-CTC (Common Terminology Criteria) v.3 criteria; CBC (complete blood count) with differential white cell and platelet counts; Serum sodium, potassium, chloride, bicarbonate, AST, ALT, alkaline phosphatase, total bilirubin, blood urea nitrogen, creatinine, and albumin; Serum CA 19-9
Time Frame: First day of each cycle
Measure: Count of Participants; unit: Participants
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 20
Participants
  diarrhea | 3
  fatigue | 5
  infection | 1
  nausea | 7
  neutrophil | 4
  pain | 5
  platelet | 1
  stomach mucostis | 1
  vomiting | 4
  wbc | 2
  other toxicity | 4

8. Secondary Outcome: pAKT (Pichia Anomala Killer Toxin) and NF (Nuclear Factor)-kappaB Activation
Description: Tumor tissue collected from paraffin
Time Frame: At start of study
Population: Data not collected
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Novasoy®, Gemcitabine & Erlotinib
Serious Adverse Events (participants affected / at risk) | 14/20
Other Adverse Events (participants affected / at risk) | 15/20
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novasoy®, Gemcitabine & Erlotinib (N=20)
Diarrhea (Gastrointestinal disorders) | 3 (3)
Fatigue (General disorders) | 5 (5)
Infection (Infections and infestations) | 1 (1)
Nausea (Gastrointestinal disorders) | 7 (7)
Neutrophil (Investigations) | 4 (4)
Pain (General disorders) | 5 (5)
Platelet (Investigations) | 1 (1)
Stomach, mucostis (Gastrointestinal disorders) | 1 (1)
White blood count (WBC) (Blood and lymphatic system disorders) | 2 (2)
Vomiting (Gastrointestinal disorders) | 4 (4)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Novasoy®, Gemcitabine & Erlotinib (N=20)
Diarrhea (Gastrointestinal disorders) | 11 (11)
Fatigue (General disorders) | 8 (8)
Hemoglobin (Blood and lymphatic system disorders) | 15 (15)
Pain (General disorders) | 7 (7)
Platelet (Investigations) | 15 (15)
Skin rash (Skin and subcutaneous tissue disorders) | 15 (15)
Stomach, mucositis (Gastrointestinal disorders) | 4 (4)
Vomiting (Gastrointestinal disorders) | 4 (4)
Neutrophil (Blood and lymphatic system disorders) | 7 (7)
WBC (white blood count) (Blood and lymphatic system disorders) | 7 (7)
Nausea (Gastrointestinal disorders) | 6 (6)

LIMITATIONS AND CAVEATS:
This study was stopped early due to the lack of efficacy.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No